CLINICAL TRIAL: NCT06243874
Title: Comparison of Greater Occipital Nerve Blockade and Sphenopalatine Ganglion Blockade in Patients With Episodic Migraine
Brief Title: Comparison of Occipital Nerve and Sphenopalatine Ganglion Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hanzade Aybuke Unal, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/381
Record Dates: First submitted 2024-01-17; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Migraine
Keywords: pain; migraine; nerve block
MeSH Terms: conditions — Migraine Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- greater occipital nerve block (Active Comparator): Following intravenous access and monitoring, participants are placed in the prone position. The medial 1/3 of the line between the protuberance occipital externa and the mastoid process is palpated. The intervention area is cleaned with antiseptic solution. Then, 2 cc of 2% lidocaine is injected into the palpated area after confirming that it is not in the vascular area by negative aspiration. Participants are observed for 30 minutes for possible complications.
  The participant will receive a block once a week for the first month and then once a month for the next 2 months.
  Interventions: Procedure: greater occipital nerve block
- transnasal sphenopalatine ganglion block (Other): Following intravenous access and monitoring, patients are placed in the supine position. A cotton swab impregnated with 2 cc of 2% lidocaine is advanced from the nostril along the upper edge of the middle turbinate until it reaches the posterior wall of the nasopharynx. The stick impregnated with local anesthetic is kept in the target area for 20 minutes. Participants are observed for 30 minutes for possible complications.
  The participant will receive a block once a week for the first month and then once a month for the next 2 months.
  Interventions: Procedure: transnasal sphenopalatine ganglion block

INTERVENTIONS:
Procedure: greater occipital nerve block — greater occipital nerve block
  Arms: greater occipital nerve block
Procedure: transnasal sphenopalatine ganglion block — transnasal sphenopalatine ganglion block
  Arms: transnasal sphenopalatine ganglion block

SUMMARY:
Migraine is a chronic disorder that causes disability. Episodic migraine can be managed by prophylactic medical treatment or interventional pain procedures. Interventional methods used in migraine treatment are greater occipital nerve blockade, lesser occipital nerve blockade, supraorbital nerve blockade, infraorbital nerve blockade, sphenopalatine ganglion blockade, botulinum toxin injection and various radiofrequency applications. The effectiveness of greater occipital nerve blockade and transnasal sphenopalatine ganglion blockade in the treatment of migraine has been proven in various studies.We aimed to evaluate the effects of repetitive greater occipital nerve blockade and transnasal sphenopalatine ganglion blockade in patients with episodic migraine.

DETAILED DESCRIPTION:
Migraine is a common primary headache and causes a significant personal, social and financial burden. Migraine is characterized by a semi-headache lasting 4-72 hours, accompanied by nausea/vomiting and photophobia/phonophobia. Migraine can be episodic or chronic. Non-steroidal anti-inflammatory drugs, triptan and ergotamine derivatives can be used in the treatment of acute migraine attacks. Beta-blockers, calcium channel blockers, antiepileptic drugs and antidepressant drugs are among the prophylactic medical treatments. When medical treatment cannot provide adequate pain palliation, in case of side effects or when the patient does not prefer medical treatment, interventional methods come to the fore. Interventional methods that applied in migraine treatment are greater occipital nerve blockade, lesser occipital nerve blockade, supraorbital nerve blockade, infraorbital nerve blockade, sphenopalatine ganglion blockade, botulinum toxin injection and various radiofrequency applications. The effectiveness of greater occipital nerve blockade and transnasal sphenopalatine ganglion blockade in the treatment of migraine has been proven in various studies.

It is stated that sphenopalatine ganglion blockade reduces the number of headache days and is effective in the treatment of acute migraine attacks. Although there are studies on the effectiveness of greater occipital nerve blockade and transnasal sphenopalatine ganglion blockade in migraine treatment, there are no studies comparing their superiority over each other. This study aims to evaluate the effects of repetitive greater occipital nerve blockade and transnasal sphenopalatine ganglion blockade on headache severity, number of days with headache, headache duration, functionality and medication use in patients with episodic migraine, and to compare whether they are superior to each other.

In this single center randomised study participants' episodic migraine will be diagnosed according to the International Classification of Headache Disorders 3rd version (ICHD-3) criteria. Demographic information of the patients, including age, gender, comorbidities, educational status, marital status and migraine duration, will be recorded. Pain intensity of patients will be evaluated using the Numeric Rating Scala (NRS 11) scale, and functionality will be evaluated using MIDAS. Before the procedure, the number of headache days in a 1-month period, headache severity, duration, amount of medication use (non-steroidal anti-inflammatory analgesic, triptan) and MIDAS score will be recorded. Participants will be randomized into 2 groups. When 21 participants are randomized in each group, participant 26 will be excluded from the list because it is in both groups. Group 1 greater occipital nerve block; It will be applied for participants 37, 27, 35, 13, 36, 18, 34, 33, 6, 12, 3, 25, 19, 1, 14, 9, 21, 38, 10, 2. Group 2 sphenopalatine block; It will be applied to patients 22, 1, 24, 11, 35, 33, 17, 14, 8, 31, 39, 5, 2, 28, 41, 36, 15, 7, 34, 27. Greater occipital nerve block will be applied to participant number 26 by repeating the procedure order since the number of participants in each group is equally divided.

Participants will receive greater occipital nerve blockade and transnasal sphenopalatine ganglion blockade once a week for the first month and then once a week for a further 1 month. At the 1st month, 2nd month and 3rd month follow-up visits of the participants, the number of headache days, average pain intensity and pain duration, MIDAS scores and the amount of medication used (non-steroidal anti-inflammatory analgesic, triptan) will be recorded with pain diaries. Participants' pain diaries, MIDAS scores and the amount of medication they use will be recorded. Additionally, possible complications in patients will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65
* Diagnosing migraine according to the International Classification of Headache Disorders 3rd version (ICHD-3) criteria
* Patients diagnosed with episodic migraine
* Failure to provide pain palliation with at least 1 prophylactic medication

Exclusion Criteria:

* Presence of psychiatric disease that is unstable/not controlled by medical treatment
* Pregnant patients
* Those with bleeding diathesis
* Patients who are allergic to local anesthetics given during the procedure
* Patients with open skull defects who have undergone craniotomy
* Patients with previous nasal/sinus surgery
* Patients with medication overuse headaches
* Presence of causes such as hypertension, vasculitis, malignancy, etc. that may cause headaches
* Patients who have received interventional headache treatment in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Post treatment 3 months
  Range pain severity 0-10, 0: No pain, 10: Worst Pain
Migraine attack duration | Post treatment 3 months
  mean migraine attack duration (hours) that patients suffer in a month.
Number of migraine days | Post treatment 3 months
  Number of migraine days that patients suffer in a month.

SECONDARY OUTCOMES:
Migraine Disability Assessment (MIDAS) questionnaire | Post treatment 3 months
  Four point likert for every question. Scores ranging from 0 to 5, little or no disability; Scores ranging from 6 to 10 indicate mild disability; Scores ranging from 11 to 20 indicate moderate disability; 21 or over, severe disability.
medication use | Post treatment 3 months
  use of medication (non-steroidal anti-inflammatory analgesic, triptan) recorded during 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanzade A Unal, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marmura MJ, Silberstein SD, Schwedt TJ. The acute treatment of migraine in adults: the american headache society evidence assessment of migraine pharmacotherapies. Headache. 2015 Jan;55(1):3-20. doi: 10.1111/head.12499. PMID 25600718
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Cady RK, Saper J, Dexter K, Cady RJ, Manley HR. Long-term efficacy of a double-blind, placebo-controlled, randomized study for repetitive sphenopalatine blockade with bupivacaine vs. saline with the Tx360 device for treatment of chronic migraine. Headache. 2015 Apr;55(4):529-42. doi: 10.1111/head.12546. Epub 2015 Mar 31. PMID 25828648
- [Background] Binfalah M, Alghawi E, Shosha E, Alhilly A, Bakhiet M. Sphenopalatine Ganglion Block for the Treatment of Acute Migraine Headache. Pain Res Treat. 2018 May 7;2018:2516953. doi: 10.1155/2018/2516953. eCollection 2018. PMID 29862074
- [Background] Malekian N, Bastani PB, Oveisgharan S, Nabaei G, Abdi S. Preventive effect of greater occipital nerve block on patients with episodic migraine: A randomized double-blind placebo-controlled clinical trial. Cephalalgia. 2022 May;42(6):481-489. doi: 10.1177/03331024211058182. Epub 2021 Nov 17. PMID 34786992
- [Derived] Unal HA, Basari A, Celiker OS, Cakar Turhan KS, Asik I, Ozgencil GE. Comparison of Greater Occipital Nerve Blockade and Sphenopalatine Ganglion Blockade in Patients with Episodic Migraine. J Clin Med. 2024 May 21;13(11):3027. doi: 10.3390/jcm13113027. PMID 38892738